CLINICAL TRIAL: NCT07040982
Title: Pilot Study of Asciminib as a Maintenance Treatment Post Cellular Therapies in Adults With Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Brief Title: Asciminib as Maintenance Treatment After Cellular Therapies for Adults With Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25023; NCI-2025-04103 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25023 (Other: City of Hope Medical center); P30CA033572 (NIH)
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1
MeSH Terms: interventions — asciminib; Specimen Handling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Asciminib) (Experimental): Patients receive asciminib PO QD or BID on days 1-28 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography during screening and as clinically indicated, and bone marrow biopsy, bone marrow aspirate and blood sample collection throughout the study.
  Interventions: Drug: Asciminib; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Other: Survey Administration

INTERVENTIONS:
Drug: Asciminib — Given PO
  Other Names: ABL 001; ABL-001; ABL001
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I trial tests the safety, side effects and best dose of asciminib as maintenance treatment for adults with Philadelphia chromosome positive acute lymphoblastic leukemia (ALL) who have undergone cellular therapies such as hematopoietic stem cell transplantation (HSCT) or chimeric antigen receptor (CAR) T cell therapy. Maintenance treatment is given to help keep cancer from coming back after it has disappeared following initial therapy. Asciminib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving asciminib may be safe and tolerable as maintenance treatment for adult patients with Philadelphia chromosome positive ALL who have undergone cellular therapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of asciminib maintenance in adults with Philadelphia chromosome (Ph)+ acute lymphoblastic leukemia (ALL) in morphological complete remission (CR) post hematopoietic stem cell transplantation (HSCT; Arm 1) or chimeric antigen receptor (CAR) T cell therapy (Arm 2).

II. Determine the recommended phase 2 dosing (RP2D) of asciminib maintenance post cellular therapies in Ph+ ALL in each arm.

SECONDARY OBJECTIVES:

I. Evaluate feasibility of asciminib maintenance measured as the number of patients who continue asciminib > 3 cycles post cellular therapy.

II. Duration of response. III. Timing for minimal residual disease (MRD) and full relapse. IV. Relapse free survival at 1 year post cellular therapy. V. Overall survival at 1 year post cellular therapy. VI. Non-relapse mortality at 1 year post cellular therapy. VII. Relapse at 1 year post cellular therapy. VIII. Rates of asciminib discontinuation and interruption due to toxicity at 1 year post cellular therapy.

IX. Rate of switching to another tyrosine kinase inhibitor (TKI) at 1 year post cellular therapy X. Rate and grade of acute graft-versus-host disease (GVHD) at 180 days post initiation of asciminib maintenance post HSCT. (Arm 1) XI. Rate and grade of chronic GVHD at 1 year post initiation of asciminib maintenance post HSCT. (Arm 1) XII. GVHD-free, relapse-free survival (GRFS) at 1 year post HSCT. (Arm 1)

EXPLORATORY OBJECTIVES:

I. For patients who are MRD-negative, evaluate MRD relapse by clonoSEQ during therapy.

II. Evaluate immune cell populations and immune reconstitution post-transplant during asciminib therapy.

III. Evaluate the impact of prevalent BCR-ABL mutations and treatment emergent BCR-ABL mutations.

IV. Evaluate B-cell aplasia and CAR T cell persistence during asciminib therapy. (Arm 2) V. Quality of life assessments using Patient Reported Outcomes Measurement Information System (PROMIS).

OUTLINE: This is a dose-escalation study of asciminib followed by a dose-expansion study.

Patients receive asciminib orally (PO) once daily (QD) or twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography during screening and as clinically indicated, and bone marrow biopsy, bone marrow aspirate and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* PRE-SCREENING: Documented informed consent of the participant and/or legally authorized representative
* PRE-SCREENING: Age ≥ 18 years
* PRE-SCREENING: Participant was diagnosed with Ph+ ALL according to World Health Organization criteria. The BCR::ABL1 translocation may be detected by fluorescence in situ hybridization (FISH), polymerase chain reaction (PCR), next generation sequencing (NGS), or cytogenetics at least once any time prior to cellular therapy. Participants may have p190 or p220 isoform, and participants with T315I mutation are not excluded
* PRE-SCREENING: Participant meets one of the following criteria:

  * Arm 1: Have a date for HSCT scheduled within the next 30 days or have received HSCT within the last 30 days. Note: all HSCT donors, conditioning regimens, and GVHD prophylaxis regimens will be acceptable.
  * Arm 2: Have a date for CAR T cell infusion scheduled within the next 30 days or have received CAR T cell infusion within the last 30 days
* PRE-SCREENING: History of pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
* PRE-SCREENING: History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Eastern Cooperative Oncology Group (ECOG) ≤ 2
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Participant is between day +30 and +150 after one of the following cellular therapies:

  * Arm 1: HSCT

    * Participants on Arm 1 must be fully engrafted post-HSCT.
  * Arm 2: CD19-targeted CAR T cell therapy (brexucabtagene autoleucel, tisagenlecleucel, obecabtagene autoleucel, investigational CD19 CAR T cell therapy)

    * Participants on Arm 2 must be fully recovered from cytopenia
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Day 30 (+/- 5 days) marrow post cellular therapy should show evidence of complete morphologic remission defined as < 5% bone marrow (BM) blasts, no extramedullary disease, and transfusion independence
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Participant should have no morphological evidence of relapse
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Absolute neutrophil count (ANC) ≥ 500/mm^3 for 3 days

  * NOTE: Patients are allowed growth factors
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Platelets ≥ 75,000/mm^3
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Hemoglobin ≥ 9g/dL
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Total bilirubin ≤ 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease)
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Aspartate aminotransferase (AST) ≤ 3.0 x ULN
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Alanine aminotransferase (ALT) ≤ 3.0 x ULN
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: serum creatinine <1.5 mg/dL
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Left ventricular ejection fraction (LVEF) ≥ 50%

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Bazett's corrected QT interval (QTcB) ≤ 480 ms

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Oxygen (O2) saturation > 90% on room air
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Seronegative for HIV antigen (Ag)/antibody (Ab) combination (combo), hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative) OR

  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* PATIENTS AFTER DAY +30 FOLLOWING CELLULAR THERAPY: Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 120 days after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior treatment failure with asciminib
* Treatment with strong inducers of CYP3A is not allowed and should be switched to an alternative at least 1 week prior to the start of study treatment
* ARM 1: Treatment with prior HSCT is allowed
* ARM 2: Treatment with prior CAR T cell therapy is allowed
* Cardiac or cardiac repolarization abnormality, including any of the following:

  * History within 6 months prior to starting study treatment of myocardial infarction (MI), or coronary artery bypass graft (CABG)
  * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third-degree AV block)
  * Fridericia's corrected QT interval (QTcF) at screening ≥ 450 msec (male patients), ≥ 470 msec (female patients)
  * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome
* History of pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
* ARM 1: Active grade 3 or higher graft-versus-host disease (GVHD) after allogeneic HSCT within 14 days of enrollment. Note: prednisone administration (flat dose of 0.5 mg/kg) is allowed. Patients receiving any other medication to control active/progressive GVHD will be excluded
* Clinically significant uncontrolled illness
* Active infection not responding to treatment
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-06-13 (Estimated); Study Completion 2028-06-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From start of treatment on day 1 to the end of cycle 1 on day 28
  Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The toxicity/adverse event information recorded on each subject will include type, severity, duration, attribution/ association with the study agent by arm and cycle. Tables will be constructed to summarize the observed incidence, severity and type of toxicity, including infection. Point estimates and 90% confidence intervals will be provided.

SECONDARY OUTCOMES:
Number of patients who have completed at least 3 cycles of asciminib and have taken ≥ 70% planned doses in each cycle post cellular therapy | Up to completion of 3 cycles (cycle length= 28 days)
  The protocol therapy will be deemed feasible if > 70% or higher of patients meet this feasibility criteria. Point estimates and 90% confidence intervals will be provided.
Duration of remission | Up to 1 year after completion of study treatment
  Point estimates and 90% confidence intervals will be provided.
Relapse including minimal residual disease (MRD) relapsed | Up to 1 year after completion of study treatment
  MRD relapse assed by polymerase chain reaction (PCR) and flow cytometry. MRD relapse is defined as detectable leukemic cells at > 0.01% in morphological remission bone marrow. However, due to rate of false positivity of PCR BCR::ABL1, confirmation is required by either positive MRD flow or/and clonoSEQ > 0.01%. Will be calculated using the competing risk method. Point estimates and 90% confidence intervals will be provided.
Relapse free survival | From start of protocol therapy to relapse, or death, up to 1 year after completion of study treatment
  Kaplan-Meier curves will be used for survival endpoints. Point estimates and 90% confidence intervals will be provided.
Overall survival | From start of protocol therapy to death regardless of cause, up to 1 year after completion of study treatment
  Kaplan-Meier curves will be used for survival endpoints. Point estimates and 90% confidence intervals will be provided.
Non-relapse mortality | From start of protocol therapy to death without relapse/progression, up to 1 year after completion of study treatment
  Will be calculated using the competing risk method. Point estimates and 90% confidence intervals will be provided.
Switching tyrosine kinase inhibitors (TKI) | Up to 1 year after completion of study treatment
  Defined as changing treatment to a different TKI due to asciminib toxicity or intolerability per the treating physician judgment. Point estimates and 90% confidence intervals will be provided.
Asciminib discontinuation | Up to 1 year
  Discontinuation is defined as not taking asciminib > 28 days due to treatment-related toxicity. Point estimates and 90% confidence intervals will be provided.
Asciminib interruption | Up to 1 year
  Interruption is defined as not taking asciminib for > 7 days because of treatment-related toxicity. Point estimates and 90% confidence intervals will be provided.
Rate of acute graft versus host disease (aGVHD) of grades 2-4 (arm 1) | From hematopoietic stem cell transplantation (HSCT) to day 180 post HSCT
  Documented/biopsy proven aGVHD is graded according to Mount Sinai Acute graft versus host disease (GVHD) International Consortium (MAGIC) grading. Point estimates and 90% confidence intervals will be provided.
Rate of aGVHD of grades 3-4 (Arm 1) | From HSCT to day 180 post HSCT
  Documented/biopsy proven aGVHD is graded according to MAGIC Grading. Point estimates and 90% confidence intervals will be provided.
GVHD-free, relapse-free survival (Arm 1) | From start of protocol therapy to the first observation of developing grade 3-4 aGVHD, chronic (c) GVHD requiring systemic therapy, relapse/progression, or death, whichever comes first, up to 1 year after completion of study treatment
  Kaplan-Meier curves will be used for survival endpoints. Point estimates and 90% confidence intervals will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Aldoss, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical center, Duarte, California, United States